CLINICAL TRIAL: NCT06728618
Title: A Single-Arm, Prospective Phase II Clinical Study on the Neoadjuvant Tislelizumab -Cetuximab - TP(cisplatin and Albumin-paclitaxel) Followed by Salvage Surgery and Adjuvant Tislelizumab -Cetuximab for Resectable, Locally Recurrent Oral and Oropharyngeal Squamous Cell Carcinoma
Brief Title: Preoperative Tislelizumab -Cetuximab - Chemotherapy Followed by Salvage Surgery and Adjuvant Tislelizumab -Cetuximab for Resectable, Locally Recurrent Oral and Oropharyngeal Squamous Cell Carcinoma
Acronym: OSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-369R2
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC); Oropharyngeal Squamous Cell Carcinoma (SCC); Resectable Oral and Oropharyngeal Squamous Cell Carcinoma; Recurrent Oral and Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; Cetuximab; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Neoadjuvant Treatment + Salvage Surgery + Adjuvant Treatment (Experimental): Neoadjuvant treatment: The participants will receive 2 cycles of combination therapy (Tislelizumab, Cetuximab, Cisplatin and Nab-paclitaxel).
  Salvage surgery: Primary tumor resection and/or lymph node dissection surgery 3-6 weeks from cycle 2 day 1.
  Adjuvant treatment: 3-8 weeks post-surgery and upto a total of half a year. The participants will receive Tislelizumab (q3w) and Cetuximab (q2w) therapy.
  Interventions:
  Drug: Tislelizumab, Cetuximab, Cisplatin and Nab-paclitaxel
  Interventions: Drug: Drug: Tislelizumab, Cetuximab, Cisplatin and Nab-paclitaxel

INTERVENTIONS:
Drug: Drug: Tislelizumab, Cetuximab, Cisplatin and Nab-paclitaxel — Neoadjuvant treatment: the participants will receive Tislelizumab 200 mg, Cisplatin 75 mg/m2, Nab-paclitaxel 260 mg/m2 (each 3-week cycle) and Cetuximab (400 mg/m2 first time and followed 250 mg/m2, day 1, day 8, day 15) for 2 cycles.
  Adjuvant treatment: the participants will receive Tislelizumab 200 mg (each 3-week cycle, a total of 8 cycle) and Cetuximab (250 mg/m2, each 2-week, a total of 12 cycle) for a total of half a year.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the combination therapy of immunotherapy (Tislelizumab), targeted therapy (Cetuximab), with chemotherapy (Cisplatin and Nab-paclitaxel) as a possible treatment before and after salvage surgery for locally recurrent oral/pharyngeal squamous cell carcinoma. The combination of Tislelizumab，Cetuximab, Cisplatin and Nab-paclitaxel will be given prior to your surgery, while Tislelizumab and Cetuximab will be continued for approximately half a year after surgery.

DETAILED DESCRIPTION:
Despite multimodality curative approaches to treat patients with oral/oropharyngeal squamous cell carcinoma (OSCC), approximately 30-40% of patients recur locally. Recurrent OSCC contributes to significant morbidity and portends overall poor survival, reflecting a situation that is difficult to treat owing to the effects of prior therapy (surgery, radiation, and/or chemotherapy) on the delicate structures of the head and neck. Both the NCCN and the CSCO head and neck cancer treatment guidelines recommend salvage surgery as a Grade I recommended curative treatment method whenever possible, as this has been shown to have a significantly better outcome as compared to patients treated non-surgically with radiation therapy with or without concurrent chemotherapy. However, salvage surgery is extremely challenging due to delicate structures of the head and neck.

Previous studies have recommended that the combination of targeted therapy (cetuximab) and chemotherapy (cisplatin, paclitaxel) has effective anti-tumor effects for recurrent/metastatic head and neck squamous cell carcinoma. Recently, newer approaches also have shown favorable safety and evidence of pathologic response when using immune-checkpoint inhibitors as neoadjuvant therapy prior to upfront, curative-intent surgery in resectable head and neck cancer. Immunotherapy is expected to be more effective with smaller amounts of disease and application of therapy when disease burden is minimal is expected to yield improved outcomes. Locally recurrent patients undergoing salvage therapy are understudied and deserves further exploration.

This is a prospective, open label, single arm, phase II, single center interventional study of neoadjuvant combination therapy of immunotherapy (Tislelizumab), targeted therapy (cetuximab), with chemotherapy (cisplatin and nab-paclitaxel) followed by salvage surgery and followed by adjuvant immunotherapy (Tislelizumab), targeted therapy (cetuximab) in patients with resectable recurrent oral/oropharyngeal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed locoregionally recurrent oral/oropharyngeal squamous cell carcinoma (including tongue, lips, gums, cheeks, floor of mouth, hard palate, soft palate, posterior molar area, lateral pharyngeal wall, posterior pharyngeal wall, tonsils).
2. Participants must have documented time of ≥ 16 weeks from completion of prior curative intent treatment for OSCC (surgery and/or radiation therapy with/without platinum chemotherapy or cetuximab targeted therapy) to diagnosis of local or locoregional recurrence.
3. Age ranges from 18 to 75 years old
4. ECOG performance status 0 or 1.
5. Expected survival ≥ 12 weeks.
6. The participants are clinically evaluated to be eligible for salvage surgery and must be intended to undergo salvage surgery.
7. There must be at least one clinically assessable lesion according to the RECIST V1.1 criteria prior to treatment.
8. The participants may have any human papillomavirus (HPV) status of the tumor. Patients with oropharyngeal cancer need to undergo HPV testing, including p16 immunohistochemistry and/or confirmatory HPV polymerase chain reaction (PCR) or in situ hybridization (ISH) testing.
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and continue contraception for 12 months after the end of treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Participants must have adequate organ and marrow function as defined below: The function of important organs meets the following requirements: (1) normal bone marrow reserve function, white blood cell (WBC) ≥ 3.0 × 10 ^ 9/L; Neutrophil count (NEUT) ≥ 1.5 × 10 ^ 9/L, platelet count (PLT) ≥ 100 × 10 ^ 9/L, hemoglobin (Hb) ≥ 90 g/L; (2) Normal renal function or serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥ 50 ml/min (Cockcroft Gault formula); (3) Normal liver function or total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); AST or ALT levels ≤ 3 times the upper limit of normal (ULN); (4) Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously. If FT3 and FT4 levels are normal, they can be included in the group).
11. The participants voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Has known distant metastasis of the disease.
2. Has received chemotherapy or radiotherapy for curative treatment of oral/oropharyngeal squamous cell carcinoma within the 16 weeks prior to enrollment in the study.
3. Has received therapy treatment with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, or anti-CTLA-4 antibody (or any other antibody acting on T cell co stimulatory or checkpoint pathways).
4. Has received live or attenuated vaccines within 30 days prior to the first dose of Tislelizumab, inactivated vaccines are allowed.
5. Has received immunosuppressive drugs within 14 days prior to the first dose of study drug, nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e. not exceeding 10 mg/day of prednisolone or other corticosteroids of equivalent physiological doses) are allowed.
6. Has an active infection that requires systematic treatment; Has a history of non -infectious pneumonia/interstitial lung disease requiring steroid treatment, or current pneumonia/interstitial lung disease; Has a known history of hepatitis B (defined as positive for hepatitis B surface antigen [HBsAg]) or known history of active hepatitis C virus (defined as detection of HCV RNA [qualitative]) infection; Has a known history of human immunodeficiency virus (HIV) infection.
7. Has received allogeneic tissue/solid organ transplantation.
8. Has not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 2) with the exception of alopecia.
9. Has obvious cardiovascular abnormalities (such as myocardial infarction, superior vena cava syndrome, and heart disease grade 2 or above diagnosed according to the New York Heart Association (NYHA) classification criteria within 3 months prior to the enrollment)。
10. Has severe clinical infection (>NCI-CTCAE 5.0 Level 2 infection);
11. Has uncontrollable hypertension (systolic blood pressure>150mmHg and/or diastolic blood pressure>90mmHg after treatment with antihypertensive drugs) or clinically significant cardiovascular diseases - such as cerebrovascular accidents (≤ 6 months before enrollment), myocardial infarction (≤ 6 months before enrollment), unstable angina, congestive heart failure classified as Grade II or above by the New York Heart Association (NYHA), or severe arrhythmias that cannot be controlled with medication or have potential impact on experimental treatment.
12. Pregnant women are not allowed to participate. Breast-feeding women who participate in this study should stop breast-feeding.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Has participated in other clinical studies within 30 days prior to enrollment.
15. Other situations that researchers consider unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Pathological Response (mPR) | 2 months
  Major pathologic response (mPR) is defined as having ≤ 10% invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes as assessed by pathologists. Rate is the proportion of treated participants who experienced mPR

SECONDARY OUTCOMES:
Rate of Pathologic complete response (PCR) | 2 months
  Pathologic complete response (PCR) is defined as having no invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes as assessed by pathologists. Rate is the proportion of treated participants who experienced PCR.
1 year Event-free Survival (EFS) Rate | 12 months
  EFS is the time from the date of study entry to the date of first record of disease progression as defined by RECIST 1.1
2 year Event-free Survival (EFS) Rate | 24 months
  EFS is the time from the date of study entry to the date of first record of disease progression as defined by RECIST 1.1
1 year Overall Survival (OS) Rate | 12 months
  OS is the time from study entry to death due to any cause
2 year Overall Survival (OS) Rate | 24 months
  OS is the time from study entry to death due to any cause
Adverse Events (AEs) | 24 months
  Number of participants experiencing any sign, symptom, disease, or worsening of preexisting conditions temporally associated with the experimental interventions or irrespective of the experimental interventions

OTHER OUTCOMES:
Changes in the Level of biomarkers for predicting therapeutic efficacy | 24 months
  Changes in the Level of PD-L1 expression, tumor mutation burden, microsatellite instability, immune cell invasion

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No